CLINICAL TRIAL: NCT00741091
Title: A Carotid Stenting Boston Scientific Surveillance Program Carotid WALLSTENT Monorail Endoprosthesis FilterWire EZ™ Embolic Protection System
Brief Title: A Carotid Stenting Boston Scientific Surveillance Program
Acronym: CABANA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2029
Record Dates: First submitted 2008-08-25; First posted 2008-08-26 (Estimated); Results first posted 2011-08-19 (Estimated); Last update posted 2011-08-24 (Estimated); Status verified 2011-08

CONDITIONS: Carotid Artery Disease
Keywords: Cerebrovascular Disease; Carotid Stent; Stent; Carotid Endarterectomy (CEA)
MeSH Terms: conditions — Carotid Artery Diseases; Cerebrovascular Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Registry (Experimental): Registry to gather data on early clinical outcomes for the Carotid WALLSTENT Endoprosthesis and FilterWire EZ System in routine clinical practice.
  Interventions: Device: Carotid WALLSTENT Monorail Endoprosthesis; Device: FilterWire EZ™ System™

INTERVENTIONS:
Device: Carotid WALLSTENT Monorail Endoprosthesis — A carotid artery stent for use in subjects at high risk for adverse events from Carotid endarterectomy (CEA) due to either anatomic or comorbid conditions who require carotid revascularization in the treatment of ipsilateral or bilateral carotid artery disease.
Device: FilterWire EZ™ System™ — Embolic protection device used in conjunction with the Carotid WALLSTENT Endoprosthesis.

SUMMARY:
CABANA is a multicenter U.S. surveillance registry that will be conducted to compile early clinical outcomes data for the Carotid WALLSTENT Endoprosthesis and FilterWire EZ System in routine clinical practice and to assess the adequacy of the Boston Scientific Corporation (BSC) Carotid Stenting Training Program.

ELIGIBILITY:
Inclusion Criteria:

* Subject at high risk for adverse events from carotid endarterectomy due to either anatomic or comorbid conditions who requires carotid revascularization in the treatment of ipsilateral or bilateral carotid artery disease.
* Subject with neurological symptoms and greater than or equal to 50% stenosis of the common, internal carotid artery and/or the bifurcation by ultrasound or angiogram OR
* Subjects without neurological symptoms and greater than or equal to 80% stenosis of the common, internal carotid artery and/or the bifurcation by ultrasound or angiogram.
* Subject has a reference vessel diameter greater than or equal to 4.0 mm and less than or equal to 9.0 mm at the target lesion and a vessel diameter distal to the target lesion of greater than or equal to 3.5 mm and less than or equal to 5.5 mm as optimal "landing zone" for placement of the FilterWire EZ System.
* Subject is willing and able to comply with all follow-up requirements.
* Subject has provided a signed informed consent prior to participation in the Registry.

Exclusion Criteria:

* Patients in whom anticoagulant and/or antiplatelet therapy is contraindicated
* Patients with severe vascular tortuosity or anatomy that would preclude the safe introduction of a guide catheter, sheath, embolic protection system or stent system
* Patients with uncorrected bleeding disorders
* Lesions in the ostium of the common carotid artery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1097 (Actual)
Dates: Start 2008-12; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Grady, Ph.D, Study Director — Boston Scientific Corporation
Locations (112):
- United States (112):
  - Baptist Medical Center Princeton, Birmingham, Alabama
  - Cardiology Associates of Mobile, Fairhope, Alabama
  - St. Joseph's Hospital and Medical Center, Barrow Neurological Institute, Phoenix, Arizona
  - Southern Arizona Vascular Institute, Tucson, Arizona
  - University of Arkansas, Little Rock, Arkansas
  - Central Cardiology Medical Clinic, Bakersfield, California
  - Los Angeles Cardiology Associates, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Hoag Hospital, Newport Beach, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - Salinas Valley Memorial Healthcare System, Salinas, California
  - University of California, San Francisco, San Francisco, California
  - St. Joseph's Medical Center, Stockton, California
  - San Ramon Regional Medical Center, Walnut Creek, California
  - University of Colorado Hospital, Aurora, Colorado
  - University of Connecticut Health Center, Farmington, Connecticut
  - Waterbury Hospital, Waterbury, Connecticut
  - Christiana Care Cardiovascular Research, Newark, Delaware
  - JFK Medical Center, Atlantis, Florida
  - Delray Medical Center, Boca Raton, Florida
  - Bethesda Memorial Hospital, Boynton Beach, Florida
  - Bradenton Cardiology, Bradenton, Florida
  - Jim Moran Heart and Vascular Research Institute, Fort Lauderdale, Florida
  - University of Florida, Gainesville, Florida
  - Aventura Hospital, Hollywood, Florida
  - University of Miami Hospital, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - MediQuest Research Group Inc at Munroe Regional Medical Center, Ocala, Florida
  - Tallahassee Research Institute, Inc., Tallahassee, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - St. Joseph's Research Institute, Atlanta, Georgia
  - Vascular Surgical Associates PC, Austell, Georgia
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Peoria Radiology Research & Education Foundation, Peoria, Illinois
  - St. John's Hospital, Prairie Education and Research Cooperative, Springfield, Illinois
  - Southern Illinois University - Memorial Medical Center, Springfield, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - The Indiana Heart Hospital, Indianapolis, Indiana
  - Norton Hospital, Louisville, Kentucky
  - Physicians and Surgeons Surgical Hospital, Monroe, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Opelousas General Health Center, Opelousas, Louisiana
  - Southern Maryland Hospital Center, Clinton, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Michigan Vascular Research Center, Flint, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - Covenant Medical Center, Saginaw, Michigan
  - Great Lakes Heart and Vascular, Saint Joseph, Michigan
  - North Memorial Medical Center, Robbinsdale, Minnesota
  - Freeman Heart & Vascular Institute, Joplin, Missouri
  - St. John's Regional Medical Center, Joplin, Missouri
  - St. Joseph Medical Center, Kansas City, Missouri
  - The Cardiac Center of Creighton University, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper University Hospital, Camden, New Jersey
  - Our Lady of Lourdes Medical Center, Cherry Hill, New Jersey
  - UMDNJ-Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - St. Michael's Medical Center, Newark, New Jersey
  - Overlook Hospital, Short Hills, New Jersey
  - New Mexico Heart Institute, PA, Albuquerque, New Mexico
  - Albany Medical Center Hospital, Albany, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Kaleida Health, Buffalo, New York
  - Mercy Hospital of Buffalo, Buffalo, New York
  - St. Joseph Hospital, Liverpool, New York
  - Mount Sinai Medical Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Wake Medical Center, Raleigh, North Carolina
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - Bethesda North Hospital, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Mercy St. Vincent, Toledo, Ohio
  - University of Toledo Medical Center, Toledo, Ohio
  - Lake West Hospital, Willoughby, Ohio
  - Oregon Stroke Center, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Central PA Cardiovascular Research Institute, Harrisburg, Pennsylvania
  - Pennsylvania Hospital of the University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Pinnacle Health at Harrisburg Hospital, Wormleysburg, Pennsylvania
  - Berks Cardiologists, Ltd., Wyomissing, Pennsylvania
  - St. Mary Medical Center, Yardley, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - South Carolina Heart Center, Columbia, South Carolina
  - University Medical Center - Greenville Memorial Hospital, Greenville, South Carolina
  - Sanford USD Medical Center - Sanford Clinical Research, Sioux Falls, South Dakota
  - Erlanger Hospital, Chattanooga, Tennessee
  - Memorial Hospital, Chattanooga, Tennessee
  - Cardiovascular Associates PC, Kingsport, Tennessee
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Baptist Hospital West, Knoxville, Tennessee
  - Baptist Memorial Hospital-Memphis, Memphis, Tennessee
  - Cardiothoracic and Vascular Surgeons (CTVS), Austin, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Presbyterian Hospital of Dallas, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - St. Luke's Episcopal Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - Peripheral Vascular Associates, San Antonio, Texas
  - University of Texas Health Science Center San Antonio, San Antonio, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Swedish Medical Center, Seattle, Washington
  - St. Joseph Hospital, Tacoma, Washington
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Hopkins LN, White CJ, Foster MT, Powell RJ, Zemel G, Diaz-Cartelle J. Carotid artery stenting and patient outcomes: the CABANA surveillance study. Catheter Cardiovasc Interv. 2014 Nov 15;84(6):997-1004. doi: 10.1002/ccd.25578. Epub 2014 Jul 18. PMID 24948033
- [Derived] White CJ, Avula SB, Mintz RT, Iskander A, Chervu A, Feldman RL, Schermerhorn ML, Woo HH, Hopkins LN. Carotid artery revascularization with distal protection in high-surgical-risk patients in routine clinical practice: rationale and design of the CABANA safety surveillance program. Catheter Cardiovasc Interv. 2012 Jan 1;79(1):167-73. doi: 10.1002/ccd.23257. Epub 2011 Oct 5. PMID 21805584

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment began on 17 December 2008. Enrollment was completed on 28 September 2010.
Groups:
- Carotid WALLSTENT Endoprothesis and FilterWire EZ System: Registry to gather data on early clinical outcomes for the Carotid WALLSTENT Endoprosthesis and FilterWire EZ System in routine clinical practice.
Period: Overall Study
Arm/Group | Carotid WALLSTENT Endoprothesis and FilterWire EZ System
Started | 1097
Completed | 1040
Not Completed | 57
Not completed — Death | 13
Not completed — Lost to Follow-up | 16
Not completed — Withdrawal by Subject | 6
Not completed — Missed Visit | 22

BASELINE CHARACTERISTICS:
Arm/Group | Carotid WALLSTENT Endoprothesis and FilterWire EZ System
Number analyzed (Participants) | 1097
Age Continuous [Mean (Standard Deviation); unit: years] | 71.3 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 414
  Male | 683
Region of Enrollment [Number; unit: participants]
  United States | 1097

OUTCOME MEASURES:

1. Primary Outcome: Composite of Major Adverse Events (MAE) Defined as Center-reported and Clinical Events Committee (CEC) Adjudicated Death, Stroke, and Myocardial Infarction (MI)
Description: Number of participants who experienced a major adverse event (MAE) 0-30 days post-procedure. MAE was defined as add death, stroke, and myocardial infarction(MI).
Time Frame: 30 days
Population: All 1097 enrolled participants were considered for analysis. A total of 1025 subjects were evaluable for MAEs. Seventy two participants were not evaluable for MAEs; 32 participants were not evaluable because the follow-up occurred less than 23 days from enrollment and 40 participants did not complete the expected follow-up.
Measure: Number; unit: Participants
Arm/Group | Carotid WALLSTENT Endoprothesis and FilterWire EZ System
Number analyzed (Participants) | 1025
Participants | 47

2. Secondary Outcome: Number of Participants With Device, Procedure, and Unrelated Adverse Events (AEs)
Description: Adverse events, serious and non-serious, were reported by all study centers. Device related adverse events were defined as any adverse event related the study device as determined by the (Principal Investigator)PI. Procedure related adverse events were defined as any adverse event related the study procedure as determine by the PI. Unrelated adverse events were determined by the PI to not be related to the study device or study procedure.
Time Frame: 30 days
Measure: Number; unit: Participants
Arm/Group | Carotid WALLSTENT Endoprothesis and FilterWire EZ System
Number analyzed (Participants) | 1097
Participants
  Participants with Device Related AEs | 139
  Participants with Procedure Related AEs | 486
  Participants with Unrelated AEs | 390

3. Secondary Outcome: Target Lesion Revascularization
Description: Number of participant with any surgical or percutaneous attempt to revascularize the target lesion after the initial treatment. The target lesion was defined as the stented segment including 0.5 cm at the proximal and distal margins of the stented segment.
Time Frame: 30 days
Measure: Number; unit: Participants
Arm/Group | Carotid WALLSTENT Endoprothesis and FilterWire EZ System
Number analyzed (Participants) | 1097
Participants | 0

4. Secondary Outcome: System Technical Success
Description: System technical success included successful delivery and deployment of the FilterWire EZ System beyond the target lesion site, delivery and deployment of the Carotid WALLSTENT Endoprosthesis at the intended location, and successful retrieval of the delivery catheter and FilterWire EZ System after stent placement. System technical success rates was calculated based on the number of participants who had both the FilterWire EZ System and Carotid WALLSTENT Endoprosthesis placement attempted.
Time Frame: 30 days
Population: To be evaluable for system technical success, subjects needed to have a Carotid WALLSTENT deployment attempted.
Measure: Number; unit: Participants
Arm/Group | Carotid WALLSTENT Endoprothesis and FilterWire EZ System
Number analyzed (Participants) | 1072
Participants | 1041

5. Secondary Outcome: Device Malfunction
Description: Device Malfunction was defined as a failure of the device to meet performance specifications or otherwise perform as intended.
Time Frame: 30 days
Measure: Number; unit: Devices
Arm/Group | Carotid WALLSTENT Endoprothesis and FilterWire EZ System
Number analyzed (Participants) | 1097
Devices | 61

ADVERSE EVENTS:
Time Frame: 30-day major adverse events (MAE) are defined as all deaths, strokes, and myocardial infarctions (MIs) that occur within 0-30 days post-procedure.
Description: Patients were also evaluated for adverse events during the procedure and at hospital discharge
Arm/Group | Carotid WALLSTENT Endoprothesis and FilterWire EZ System
Serious Adverse Events (participants affected / at risk) | 230/1097
Other Adverse Events (participants affected / at risk) | 332/1097
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carotid WALLSTENT Endoprothesis and FilterWire EZ System (N=1097)
Anaemia (Blood and lymphatic system disorders) | 16 (16)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 8 (9)
Angina unstable (Cardiac disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 4 (4)
Atrial flutter (Cardiac disorders) | 2 (2)
Atrioventricular block first degree (Cardiac disorders) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 14 (14)
Cardiac arrest (Cardiac disorders) | 5 (5)
Cardiac failure (Cardiac disorders) | 3 (3)
Cardiac failure congestive (Cardiac disorders) | 7 (8)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 5 (5)
Sick sinus syndrome (Cardiac disorders) | 1 (1)
Sinus arrest (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Blindness (Eye disorders) | 1 (1)
Blindness transient (Eye disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Retinal artery occlusion (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (4)
Gastrointestinal ulcer (Gastrointestinal disorders) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5)
Oesophagitis (Gastrointestinal disorders) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1)
Vomiting (General disorders) | 2 (2)
Adverse drug reaction (General disorders) | 3 (3)
Asthenia (General disorders) | 4 (4)
Catheter site discharge (General disorders) | 2 (2)
Catheter site haematoma (General disorders) | 5 (5)
Catheter site haemorrhage (General disorders) | 1 (1)
Catheter site related reaction (General disorders) | 2 (2)
Chills (General disorders) | 1 (1)
Death (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Generalised oedema (General disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 3 (3)
Pyrexia (General disorders) | 3 (3)
Cholecystitis (Hepatobiliary disorders) | 2 (2)
Anaphylactic reaction (Immune system disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Catheter site infection (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1)
Kidney infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 7 (7)
Pneumonia bacterial (Infections and infestations) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 2 (2)
Staphylococcal infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 7 (7)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Brain herniation (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Incision site haematoma (Injury, poisoning and procedural complications) | 1 (1)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1)
Procedural hypertension (Injury, poisoning and procedural complications) | 1 (1)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (2)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2)
Blood creatinine increased (Investigations) | 2 (2)
Blood pressure increased (Investigations) | 1 (1)
Cardiac stress test abnormal (Investigations) | 1 (1)
Electrocardiogram change (Investigations) | 2 (2)
Haematocrit decreased (Investigations) | 2 (2)
Haemoglobin abnormal (Investigations) | 1 (1)
Haemoglobin decreased (Investigations) | 4 (4)
Troponin increased (Investigations) | 2 (2)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1 (1)
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung carcinoma cell type unspecified stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1)
Carotid artery occlusion (Nervous system disorders) | 1 (1)
Carotid artery thrombosis (Nervous system disorders) | 2 (3)
Cerebral artery thrombosis (Nervous system disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (2)
Cerebral infarction (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 25 (25)
Convulsion (Nervous system disorders) | 6 (6)
Dizziness (Nervous system disorders) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 3 (4)
Headache (Nervous system disorders) | 3 (3)
Hemiparesis (Nervous system disorders) | 3 (3)
Hemiplegia (Nervous system disorders) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Sensory disturbance (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Syncope vasovagal (Nervous system disorders) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 9 (9)
Tremor (Nervous system disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (2)
Delirium (Psychiatric disorders) | 1 (1)
Disorientation (Psychiatric disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 3 (3)
Haematuria (Renal and urinary disorders) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Renal failure acute (Renal and urinary disorders) | 5 (5)
Renal failure chronic (Renal and urinary disorders) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Toe amputation (Surgical and medical procedures) | 1 (1)
Aortic aneurysm (Vascular disorders) | 1 (1)
Arterial spasm (Vascular disorders) | 2 (2)
Arterial thrombosis limb (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 3 (3)
Haemorrhage (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 4 (4)
Hypotension (Vascular disorders) | 48 (48)
Iliac artery stenosis (Vascular disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 3 (4)
Peripheral vascular disorder (Vascular disorders) | 1 (2)
Shock (Vascular disorders) | 1 (1)
Temporal arteritis (Vascular disorders) | 1 (1)
Vasospasm (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carotid WALLSTENT Endoprothesis and FilterWire EZ System (N=1097)
Bradycardia (Cardiac disorders) | 94 (97)
Catheter site haematoma (General disorders) | 69 (71)
Catheter site haemorrhage (General disorders) | 57 (59)
Headache (Nervous system disorders) | 58 (59)
Hypotension (Vascular disorders) | 162 (168)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PI is that the Sponsor can review results communications prior to public release and can embargo communication regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the Sponsor for review. The Sponsor can require changes to the communication to remove any confidential information or other proprietary information of Sponsor.